CLINICAL TRIAL: NCT00003976
Title: Phase I Study to Determine the Safety of E7070 in Patients With a Solid Tumor on a Single IV Infusion Repeated Every 3 Weeks
Brief Title: E7070 in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16973; EORTC-16973; EISAI-E7070-E044-101
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: indisulam

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of E7070 in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of E7070 in patients with solid tumors. II. Assess the qualitative and quantitative toxicity in terms of predictability, duration, intensity, onset, reversibility, and dose relationship of this treatment regimen in this patient population. III. Determine a safe dose for phase II evaluation. IV. Assess the pharmacokinetics of this treatment regimen in these patients. V. Determine any possible antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive E7070 IV over 1 hour once every 3 weeks. Treatment continues for at least 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of E7070 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor not amenable to standard therapy No brain tumor involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin less than 1.5 mg/dL Transaminases and alkaline phosphatase no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN for liver metastases) Renal: Creatinine no greater than 1.4 mg/dL OR Creatinine clearance at least 60 mL/min Other: No active bacterial infections (e.g., abscess or fistula) No other nonmalignant disease that precludes protocol therapy No history of alcoholism, drug addiction, or psychotic disorders that would prevent compliance No glaucoma Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) Endocrine therapy: At least 4 weeks since prior anticancer hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy (6 weeks for extensive radiotherapy) No concurrent radiotherapy except for localized palliation Surgery: Not specified Other: No other concurrent investigational drugs or antitumor drugs No sulphonylureas or anti-arrhythmic agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Armand, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (27):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research-Brussels Branch, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland